CLINICAL TRIAL: NCT02235389
Title: A Multicentre, Feasibility Study of Pre-hospital Treatment of Acute Myocardial Infarction Based on Diagnosis by Interpretation of Remotely Acquired ECG and Thrombolysis With Accelerated Alteplase ( Actilyse®). Pre-Hospital Alteplase Remote Advice of Hospital (PHARAOH)
Brief Title: A Study of Pre-hospital Treatment of Acute Myocardial Infarction Based on Diagnosis by Interpretation of Remotely Acquired ECG and Thrombolysis With Accelerated Alteplase ( Actilyse®)
Acronym: PHARAOH
Status: Terminated | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 135.301
Record Dates: First submitted 2014-09-09; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Tissue Plasminogen Activator; Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Administration of thrombolytic treatment with PHARAOH: Pre-Hospital Alteplase Remote Advice of Hospital (PHARAOH)
  Interventions: Drug: Alteplase (Actilyse)
- Standard therapy with thrombolytic treatment in Hospital
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Alteplase (Actilyse)
  Groups: Administration of thrombolytic treatment with PHARAOH
Drug: Standard therapy
  Groups: Standard therapy with thrombolytic treatment in Hospital

SUMMARY:
The general aim of this study was to assess the feasibility of treating acute myocardial infarction (AMI) by physician-directed pre-hospital thrombosis, using accelerated alteplase (Actilyse®) and a diagnostic technique involving remote electrocardiogram (ECG) acquisition by paramedics

ELIGIBILITY:
Inclusion Criteria:

* Ischemic cardiac pain of >= 20 minutes and <= 6 hours
* Age 18 - 80 years
* Ability to give informed consent (witnessed verbal or written)
* Ability to follow protocol and comply with follow -up requirements

Exclusion Criteria:

* Current participation in another clinical trial
* Patient will be ineligible for pre hospital administration of actilyse if any of the following apply:

  * Acute myocardial infarction (AMI) treated with a thrombolytic agent within the preceding 4 days
  * BP (blood pressure) > 180/100 mmHg (on one measurement)
  * Significant bleeding disorder within the past 6 months
  * Major surgery, biopsy of a parenchymal organ, or significant trauma (including any trauma associated with the current AMI) within 3 months
  * History of stroke, transient ischaemic attack, or central nervous system structural damage (e.g. neoplasm, aneurysm, intracranial surgery)
  * Oral anticoagulation
  * Recent (within 10 days) non - compressible vascular puncture
  * Pregnancy (positive urine pregnancy test) or lactation, parturition within the previous 30 days, or female of childbearing potential not using adequate birth control (oral contraception)
  * Severe liver disease, including hepatic failure, cirrhosis portal hypertension (oesophageal varices) and active hepatitis
  * Diabetes with definite history of retinopathy
  * Other serious illness (e.g. malignancy, active infection)
  * Bacterial endocarditis / pericarditis
  * Acute pancreatitis
  * Documented ulcerative gastrointestinal disease during last 3 month, arterial aneurysms, arterial / venous malformations
  * Any other condition that the investigator feels would pose a significant hazard to the subject if the investigational therapy was to be initiated
* Patients who are not excluded from thrombolytic therapy by the criteria above will, in addition, need to satisfy the following 'inclusion' criteria prior to the pre - hospital thrombolysis:

  * 12 lead ECG criteria: ST segment elevation >= 0.1 mV in two contiguous electrocardiogram (ECG) standard leads indicative of AMI, or ST elevation >= 0.2 mV in two contiguous chest leads and all left bundle branch block (LBBB) with clinical indication of AMI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction treated by paramedics under the direction of hospital physicians
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 1998-02; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Percentage of equipment function / reliability | Up to 12 month after drug administration
Time between pre-hospital evaluation and treatment | Up to 12 month after drug administration
Percentage of acute myocardial infarction (AMI) patients, whose symptoms were recognized by paramedics | Up to 12 month after drug administration
Percentage of patients correctly diagnosed as suffering acute myocardial infarction by remote ECG interpretation | Up to 12 month after drug administration
Percentage of patients incorrectly diagnosed as suffering acute myocardial infarction by remote ECG interpretation | Up to 12 month after drug administration
Percentage of patients receiving pre- hospital thrombolysis in the absence of a subsequently confirmed diagnosis of acute myocardial infarction | Up to 12 month after drug administration
Percentage of patients giving consent to pre- hospital evaluation using remote electrocardiogram (ECG) | Up to 12 month after drug administration
Number of patients with adverse events | Up to 12 month after drug administration
Patient status at 30 days post myocardial infarction | Up to 30 days after drug administration